CLINICAL TRIAL: NCT05512936
Title: Cross-cultural Adaptation, Reliability, and Validity of the Turkish Version of Self-perceived Barriers for Physical Activity Questionnaire
Brief Title: The Turkish Version of the Self-perceived Barriers for Physical Activity Questionnaire
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tansu Birinci, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: 210822
Record Dates: First submitted 2022-08-20; First posted 2022-08-23 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2023-02

CONDITIONS: Physical Inactivity; Health Behavior; Quality of Life
Keywords: Health; Physical activity; Psychometrics; Quality of life
MeSH Terms: conditions — Sedentary Behavior; Health Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Self-perceived Barriers for Physical Activity Questionnaire (SBPAQ) is originally developed in Spanish to evaluate self-perceived barriers for physical activity participation in healthy individuals. The purpose of this study is to translate and cross-culturally adapt the SBPAQ into Turkish and investigate its psychometric properties.

DETAILED DESCRIPTION:
The Self-perceived Barriers for Physical Activity Questionnaire (SBPAQ) is originally developed in Spanish to evaluate self-perceived barriers for physical activity participation in healthy individuals. The purpose of this study is to translate and cross-culturally adapt the SBPAQ into Turkish and investigate its psychometric properties. Approximately two hundred healthy individuals aged between 18-65 years will be included. For cross-cultural adaptation, two bi-lingual translators will use the back-translation procedure. After the questionnaire will be translated into Turkish, the reliability, validity, and internal consistency of the Turkish version of SBPAQ (SBPAQ-T) will be tested. The questionnaire will be applied twice within 7 days to evaluate the test-retest reliability and to calculate the "Intraclass Correlation Coefficient" (ICC). Pearson correlation coefficient will be used to analyze construct and convergent/divergent validity. The construct validity of SBPAQ-T will be analyzed based on its correlation with the Physical Activity Barriers Questionnaire, International Physical Activity Questionnaire-Short Form, and Short Form-12. The Cronbach's Alpha will be calculated to determine internal consistency. The level of significance is considered as 0.05. The floor and ceiling effects will be detected.

ELIGIBILITY:
Inclusion Criteria:

* Being aged between 18-65 years
* Having the ability to read and write Turkish
* Having good cooperation to complete the assessment
* Being a volunteer to participate in the study

Exclusion Criteria:

* Having any musculoskeletal disease, cardiorespiratory system problem, or movement limitation in any joint that prevents participation in physical activity
* Having undergone surgery affecting the musculoskeletal system in the last 3 months
* Being pregnant
* Having a neurological or cognitive impairment
* Having any movement disorder
* Having the vision and/or hearing problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants are healthy individuals aged between 18-65 years.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-21 (Actual)

PRIMARY OUTCOMES:
The Self-perceived Barriers for Physical Activity Questionnaire (SBPAQ) | Baseline (First assessment)
  The Self-perceived Barriers for Physical Activity Questionnaire (SBPAQ) is composed of 17 items and 4 subscales: 1) Body image &psychosocial anxiety (5-item); 2) Fatigue & laziness (3-item); 3) Obligations & lack of time (3-item); and 4) Environment & facilities (4-item). The SBPAQ is a comprehensive and valid scoring system to evaluate perceived barriers to physical activity participation in healthy individuals.

SECONDARY OUTCOMES:
The Self-perceived Barriers for Physical Activity Questionnaire (SBPAQ) | Within a 7-day period after the first assessment (Second assessment)
  The Self-perceived Barriers for Physical Activity Questionnaire (SBPAQ) is composed of 17 items and 4 subscales: 1) Body image &psychosocial anxiety (5-item); 2) Fatigue & laziness (3-item); 3) Obligations & lack of time (3-item); and 4) Environment & facilities (4-item). The SBPAQ is a comprehensive and valid scoring system to evaluate perceived barriers to physical activity participation in healthy individuals.
International Physical Activity Questionnaire - Short Form (IPAQ-SF) | Baseline (First assessment)
  International Physical Activity Questionnaire - Short Form (IPAQ-SF) is composed of 7 items to assess the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in metabolic equivalent (MET)-min/week and time spent sitting in youth 15 years of age and older.
Physical Activity Barriers Questionnaire (PABQ) | Baseline (First assessment)
  Physical Activity Barriers Questionnaire (PABQ) is composed of 24 items and 3 subscales: 1) Personal Barriers (14-item); 2) Social Barriers (3-item); 3) Environmental Barriers (6-item). The PABQ is a comprehensive and valid scoring system to evaluate perceived barriers to physical activity participation in healthy individuals.
Short Form-12 (SF-12) | Baseline (First assessment)
  Short Form-12 (SF-12), which is developed based on Short Form-36, consists of 12 items: 7 items dealing with the physical components scores (PCS-12) and 5 items related to the mental components scores (MCS-12) of SF-12. Range of both scores is 0 to 100, where the higher scores indicate better health related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Tansu Birinci, PT, PhD, Principal Investigator — Istanbul Medeniyet Universitesi
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Bakırkoy, Turkey (Türkiye)